CLINICAL TRIAL: NCT04035668
Title: An Adaptive Phase 2 Randomized Double-blind, Placebo-controlled Multi-center Study to Evaluate the Safety and Efficacy of Multiple LOU064 Doses in Patients With Moderate to Severe Sjögren's Syndrome (LOUiSSe)
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of LOU064 in Patients With Moderate to Severe Sjögren's Syndrome
Acronym: LOUiSSe
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CLOU064E12201; 2018-004387-54 (EudraCT Number)
Record Dates: First submitted 2019-07-08; First posted 2019-07-29 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Sjögren Syndrome
Keywords: LOU064; remibrutinib; Sjogren Syndrome; Dry Eye Syndromes; Pathological Processes; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Xerostomia; Salivary Gland Diseases; Mouth Diseases; Stomatognathic Diseases; Lacrimal Apparatus Diseases; Eye Diseases; Connective Tissue Diseases; Autoimmune Diseases; Immune System Diseases
MeSH Terms: conditions — Sjogren's Syndrome; Dry Eye Syndromes; Pathologic Processes; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Xerostomia; Salivary Gland Diseases; Mouth Diseases; Stomatognathic Diseases; Lacrimal Apparatus Diseases; Eye Diseases; Connective Tissue Diseases; Autoimmune Diseases; Immune System Diseases | interventions — remibrutinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Remibrutinib 100 mg bid (Experimental): Remibrutinib 100 mg twice daily (bid)
  Interventions: Drug: Remibrutinib
- Remibrutinib 100 mg qd (Experimental): Remibrutinib 100 mg once daily (qd)
  Interventions: Drug: Remibrutinib; Drug: Placebo
- Placebo (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Remibrutinib — Remibrutinib 100 mg was administered orally as two 50 mg hard gelatin capsules. Patients in the remibrutinib 100 mg bid dose group took 2 capsules of active medication in the morning and 2 capsules of active medication in the evening. Patients in the remibrutinib 100 mg qd dose group took 2 capsules of active medication in the morning and 2 capsules of the placebo in the evening.
  Other Names: LOU064
  Arms: Remibrutinib 100 mg bid; Remibrutinib 100 mg qd
Drug: Placebo — Placebo was administered orally as two hard gelatin capsules. Patients in the placebo dose group took 2 capsules of placebo in the morning and 2 capsules of placebo in the evening.
  Arms: Placebo; Remibrutinib 100 mg qd

SUMMARY:
This was an adaptive design phase 2 study to establish safety and efficacy; and to characterize the dose-response of LOU064 in subjects with moderate to severe Sjögren's syndrome. LOU064 is an oral Bruton's tyrosine kinase (BTK) inhibitor.

DETAILED DESCRIPTION:
This study was planned as an adaptive Phase 2 randomized, double-blind, placebo-controlled, multi-center, integrated dose-ranging study to evaluate the safety and efficacy of multiple remibrutinib doses in patients with moderate to severe Sjögren's Syndrome.

Of the initially planned two parts, only Part 1 of the study was conducted. In Part 1, the highest expected biologically active single dose of remibrutinib (100 mg) was tested in two different dosing regimens, a once daily dose (qd) or twice daily dose (bid), and compared to the placebo group. Each patient in Part 1 of the study underwent a screening period of up to 6 weeks, a treatment period of 24 weeks, and a follow-up period of 30 days post-treatment before the End of Study (EOS) visit. The total duration for each patient in the study, including Screening, was up to 35 weeks. For the treatment period, patients were randomized in a 1:1:1 ratio to one of the 3 treatment groups: remibrutinib 100 mg bid, remibrutinib 100 mg qd and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SjS according to the 2016 ACR/EULAR criteria
* Screening ESSDAI (based on weighted score) ≥ 5 derived from 8 domains
* Screening ESSPRI ≥ 5
* Seropositive for anti-Ro/SSA antibodies at or within 3 months prior to screening
* Unstimulated salivary flow > 0 mL/min.

Exclusion Criteria:

* Sjögren's Syndrome overlap syndromes with another autoimmune disease as primary illness
* DMARDs or kinase inhibitors within 3 months prior to baseline above certain doses OR maintained during study
* Rituximab or other B cell depleting drug within 12 months of Screening .
* Current use of prednisone or equivalent > 15mg/d or dose change within 2 weeks prior to Screening
* Use of medication known to cause, as a major side effect, dry mouth / eyes
* HIV, Hepatitis C, Hepatitis B, known or suspected history of an ongoing, chronic or recurrent infectious disease such as tuberculosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (25):
- Novartis Investigative Site, Boston, Massachusetts, United States
- Australia (3):
  - Novartis Investigative Site, Woodville, South Australia
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Clayton, Victoria
- Novartis Investigative Site, Ghent, Belgium
- Novartis Investigative Site, Sofia, Bulgaria
- China (3):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Chengdu, Sichuan
- Novartis Investigative Site, Glostrup Municipality, Denmark
- Novartis Investigative Site, Berlin, Germany
- Novartis Investigative Site, Debrecen, Hungary
- Spain (5):
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Lausanne
- Taiwan (3):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
- United Kingdom (3):
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, Swindon
  - Novartis Investigative Site, Tyne and Wear

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Dorner T, Kaul M, Szanto A, Tseng JC, Papas AS, Pylvaenaeinen I, Hanser M, Abdallah N, Grioni A, Santos Da Costa A, Ferrero E, Gergely P, Hillenbrand R, Avrameas A, Cenni B, Siegel RM. Efficacy and safety of remibrutinib, a selective potent oral BTK inhibitor, in Sjogren's syndrome: results from a randomised, double-blind, placebo-controlled phase 2 trial. Ann Rheum Dis. 2024 Feb 15;83(3):360-371. doi: 10.1136/ard-2023-224691. PMID 37932009
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 26 investigative sites in 12 countries.
Pre-assignment Details: The screening period of up to 6 weeks began after the subject had provided written informed consent. Eligible subjects were randomized in a 1:1:1 ratio to one of the 3 treatment groups.
Period: Overall Study
Arm/Group | Remibrutinib 100 mg Bid | Remibrutinib 100 mg qd | Placebo
Started | 24 | 25 | 24
Completed | 17 | 17 | 21
Not Completed | 7 | 8 | 3
Not completed — Adverse Event | 3 | 4 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 2 | 1 | 1
Not completed — Subject Decision | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remibrutinib 100 mg Bid | Remibrutinib 100 mg qd | Placebo | Total
Number analyzed (Participants) | 24 | 25 | 24 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (15.21) | 54.8 (10.51) | 51.0 (13.94) | 51.8 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 23 | 71
  Male | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 7 | 7 | 7 | 21
  White | 17 | 17 | 16 | 50
  Unknown | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) Total Score at Week 24
Description: ESSDAI is a validated disease outcome measure for Sjögren's Syndrome. The instrument contains 12 organ-specific domains contributing to disease activity: constitutional, lymphadenopathy, glandular, articular, cutaneous, pulmonary, renal, muscular, peripheral nervous system, central nervous system, hematological and biological. For each domain, features of disease activity were scored according to their severity. These scores were summed across the 12 domains in a weighted manner to provide the total score. ESSDAI total score ranges from 0 to 123 with higher values indicating more disease activity. A negative change from baseline indicates improvement.
  The baseline value is defined as the last assessment performed prior to administration of the first dose of study treatment.
  A mixed effect model for repeated measurements (MMRM) was fitted to the changes from baseline in ESSDAI for all post-baseline time points up to Week 24. Values estimated from the model are presented in this table.
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set (FAS) with a valid assessment for the outcome measure. FAS included all participants who were randomized in the study.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Groups:
- Any Remibrutinib: Patients in any of the two remibrutinib treatment groups
Arm/Group | Remibrutinib 100 mg qd | Remibrutinib 100 mg Bid | Any Remibrutinib | Placebo
Number analyzed (Participants) | 24 | 24 | 48 | 24
score on scale | -4.70 (0.78) | -3.70 (0.80) | -4.20 (0.56) | -1.34 (0.74)
Statistical Analysis 1: Comparison: Any Remibrutinib vs Placebo; Test type: Superiority; p = 0.002, MMRM — one-sided p-value; Mean Difference (Final Values) = -2.86, 95% CI 2-sided [-4.71 to -1.01] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 2: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Test type: Other; MMRM; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-3.24 to 1.25] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)

2. Secondary Outcome: Change From Baseline in ESSDAI Total Score Over Time
Description: as for outcome 1
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16 and Week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Remibrutinib 100 mg qd | Remibrutinib 100 mg Bid | Any Remibrutinib | Placebo
Number analyzed (Participants) | 24 | 24 | 48 | 24
score on scale
  Week 2 | -1.68 (0.52) | -1.05 (0.52) | -1.37 (0.37) | -0.37 (0.55)
  Week 4 | -2.57 (0.60) | -2.54 (0.62) | -2.55 (0.43) | -0.79 (0.61)
  Week 8 | -2.74 (0.72) | -2.93 (0.71) | -2.83 (0.51) | -2.36 (0.69)
  Week 12 | -3.66 (0.74) | -2.56 (0.75) | -3.11 (0.53) | -1.92 (0.73)
  Week 16 | -4.02 (0.71) | -2.57 (0.74) | -3.29 (0.51) | -2.16 (0.69)
  Week 20 | -4.40 (0.73) | -3.26 (0.75) | -3.83 (0.52) | -1.84 (0.69)
Statistical Analysis 1: Comparison: Any Remibrutinib vs Placebo; Week 2; Test type: Superiority; p = 0.065, MMRM — one-sided p-value; Mean Difference (Final Values) = -0.99, 95% CI 2-sided [-2.29 to 0.30] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 2: Comparison: Any Remibrutinib vs Placebo; Week 4; Test type: Superiority; p = 0.010, MMRM — one-sided p-value; Mean Difference (Final Values) = -1.76, 95% CI 2-sided [-3.24 to -0.29] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 3: Comparison: Any Remibrutinib vs Placebo; Week 8; Test type: Superiority; p = 0.289, MMRM — one-sided p-value; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-2.17 to 1.22] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 4: Comparison: Any Remibrutinib vs Placebo; Week 12; Test type: Superiority; p = 0.093, MMRM — one-sided p-value; Mean Difference (Final Values) = -1.19, 95% CI 2-sided [-2.97 to 0.59] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 5: Comparison: Any Remibrutinib vs Placebo; Week 16; Test type: Superiority; p = 0.094, MMRM — one-sided p-value; Mean Difference (Final Values) = -1.13, 95% CI 2-sided [-2.84 to 0.57] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 6: Comparison: Any Remibrutinib vs Placebo; Week 20; Test type: Superiority; p = 0.012, MMRM — one-sided p-value; Mean Difference (Final Values) = -1.99, 95% CI 2-sided [-3.71 to -0.28]; Difference (Any remibrutinib - Placebo)
Statistical Analysis 7: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 2; Test type: Other; MMRM; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-2.10 to 0.84] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 8: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 4; Test type: Other; MMRM; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-1.75 to 1.69] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 9: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 8; Test type: Other; MMRM; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-1.83 to 2.21] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 10: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 12; Test type: Other; MMRM; Mean Difference (Final Values) = -1.10, 95% CI 2-sided [-3.20 to 1.01] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 11: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 16; Test type: Other; MMRM; Mean Difference (Final Values) = -1.45, 95% CI 2-sided [-3.50 to 0.60] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 12: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 20; Test type: Other; MMRM; Mean Difference (Final Values) = -1.14, 95% CI 2-sided [-3.22 to 0.95] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)

3. Secondary Outcome: Change From Baseline in EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) Total Score Over Time
Description: ESSPRI is an established disease outcome measure for Sjögren's Syndrome. It consists of three domains of dryness, pain, and fatigue. The patient can assess the severity of symptoms they experience on a single 0-10 numerical scale for each of the three domains. The ESSPRI score is defined as the mean of scores from the three scales: (dryness + pain +fatigue) /3. ESSPRI total score ranges from 0 to 10 with higher values indicating more disease symptoms. A negative change from baseline indicates improvement.
  The baseline value is defined as the last assessment performed prior to administration of the first dose of study treatment.
  A mixed effect model for repeated measurements (MMRM) was fitted to the changes from baseline in ESSPRI for all post-baseline time points up to Week 24. Values estimated from the model are presented in this table.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20 and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Remibrutinib 100 mg qd | Remibrutinib 100 mg Bid | Any Remibrutinib | Placebo
Number analyzed (Participants) | 24 | 24 | 48 | 24
score on scale
  Week 2 | -0.44 (0.26) | 0.18 (0.26) | -0.13 (0.18) | -0.09 (0.27)
  Week 4 | -0.72 (0.30) | -0.14 (0.30) | -0.43 (0.21) | -0.35 (0.30)
  Week 8 | -0.83 (0.31) | -0.38 (0.31) | -0.60 (0.22) | -0.57 (0.29)
  Week 12 | -0.88 (0.31) | -0.32 (0.31) | -0.60 (0.22) | -0.66 (0.29)
  Week 16 | -0.77 (0.36) | -0.39 (0.37) | -0.58 (0.26) | -0.71 (0.34)
  Week 20 | -0.92 (0.38) | -0.74 (0.39) | -0.83 (0.27) | -0.92 (0.36)
  Week 24 | -1.17 (0.34) | -0.76 (0.35) | -0.96 (0.24) | -1.13 (0.31)
Statistical Analysis 1: Comparison: Any Remibrutinib vs Placebo; Week 2; Test type: Superiority; p = 0.460, MMRM — one-sided p-value; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.69 to 0.62] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 2: Comparison: Any Remibrutinib vs Placebo; Week 4; Test type: Superiority; p = 0.418, MMRM — one-sided p-value; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.82 to 0.66] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 3: Comparison: Any Remibrutinib vs Placebo; Week 8; Test type: Superiority; p = 0.466, MMRM — one-sided p-value; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.76 to 0.70] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 4: Comparison: Any Remibrutinib vs Placebo; Week 12; Test type: Superiority; p = 0.560, MMRM — one-sided p-value; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.67 to 0.79] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 5: Comparison: Any Remibrutinib vs Placebo; Week 16; Test type: Superiority; p = 0.616, MMRM — one-sided p-value; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.73 to 0.99] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 6: Comparison: Any Remibrutinib vs Placebo; Week 20; Test type: Superiority; p = 0.581, MMRM — one-sided p-value; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.81 to 0.99]; Difference (Any remibrutinib - Placebo)
Statistical Analysis 7: Comparison: Any Remibrutinib vs Placebo; Week 24; Test type: Superiority; p = 0.663, MMRM — one-sided p-value; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.62 to 0.96] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 8: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 2; Test type: Other; MMRM; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-1.35 to 0.11] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 9: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 4; Test type: Other; MMRM; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.42 to 0.26] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 10: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 8; Test type: Other; MMRM; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-1.31 to 0.42] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 11: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 12; Test type: Other; MMRM; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-1.44 to 0.31] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 12: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 16; Test type: Other; MMRM; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-1.39 to 0.65] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 13: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 20; Test type: Other; MMRM; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-1.39 to 0.65] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 14: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 24; Test type: Other; MMRM; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-1.37 to 0.57] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)

4. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F) Total Score Over Time
Description: FACIT-F v4 is a short, 13-item, easy-to-administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue was measured on a 5-point Likert scale (0 = not at all, 1 = a little bit, 2 = somewhat, 3 = quite a bit, 4 = very much). FACIT-F total score ranges from 0 to 52 with higher values indicating higher quality of life (less fatigue). A positive change from baseline is a favorable outcome.
  The baseline value is defined as the last assessment performed prior to administration of the first dose of study treatment.
  A mixed effect model for repeated measurements (MMRM) was fitted to the changes from baseline in FACIT-F for all post-baseline time points up to Week 24. Values estimated from the model are presented in this table.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20 and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Remibrutinib 100 mg qd | Remibrutinib 100 mg Bid | Any Remibrutinib | Placebo
Number analyzed (Participants) | 24 | 23 | 47 | 23
score on scale
  Week 2 | 1.80 (1.32) | -0.51 (1.35) | 0.64 (0.95) | 3.37 (1.43)
  Week 4 | 4.83 (1.50) | 3.97 (1.57) | 4.40 (1.09) | 3.51 (1.58)
  Week 8 | 4.00 (1.64) | 3.79 (1.66) | 3.90 (1.17) | 5.26 (1.60)
  Week 12 | 4.88 (1.80) | 4.25 (1.86) | 4.56 (1.30) | 7.30 (1.77)
  Week 16 | 4.40 (1.97) | 3.29 (2.08) | 3.84 (1.44) | 7.73 (1.98)
  Week 20 | 10.01 (2.20) | 4.32 (2.30) | 7.16 (1.60) | 5.77 (2.17)
  Week 24 | 8.17 (2.45) | 4.64 (2.55) | 6.40 (1.77) | 7.45 (2.32)
Statistical Analysis 1: Comparison: Any Remibrutinib vs Placebo; Week 2; Test type: Superiority; p = 0.940, MMRM — one-sided p-value; Mean Difference (Final Values) = -2.73, 95% CI 2-sided [-6.18 to 0.73] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 2: Comparison: Any Remibrutinib vs Placebo; Week 4; Test type: Superiority; p = 0.322, MMRM — one-sided p-value; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [-2.95 to 4.74] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 3: Comparison: Any Remibrutinib vs Placebo; Week 8; Test type: Superiority; p = 0.753, MMRM — one-sided p-value; Mean Difference (Final Values) = -1.36, 95% CI 2-sided [-5.32 to 2.59] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 4: Comparison: Any Remibrutinib vs Placebo; Week 12; Test type: Superiority; p = 0.891, MMRM — one-sided p-value; Mean Difference (Final Values) = -2.74, 95% CI 2-sided [-7.13 to 1.66] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 5: Comparison: Any Remibrutinib vs Placebo; Week 16; Test type: Superiority; p = 0.941, MMRM — one-sided p-value; Mean Difference (Final Values) = -3.88, 95% CI 2-sided [-8.77 to 1.01] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 6: Comparison: Any Remibrutinib vs Placebo; Week 20; Test type: Superiority; p = 0.304, MMRM — one-sided p-value; Mean Difference (Final Values) = 1.39, 95% CI 2-sided [-4.01 to 6.79]; Difference (Any remibrutinib - Placebo)
Statistical Analysis 7: Comparison: Any Remibrutinib vs Placebo; Week 24; Test type: Superiority; p = 0.640, MMRM — one-sided p-value; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-6.89 to 4.79] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 8: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 2; Test type: Other; MMRM; Mean Difference (Final Values) = 2.32, 95% CI 2-sided [-1.44 to 6.07] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 9: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 4; Test type: Other; MMRM; Mean Difference (Final Values) = 0.86, 95% CI 2-sided [-3.46 to 5.18] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 10: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 8; Test type: Other; MMRM; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-4.43 to 4.83] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 11: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 12; Test type: Other; MMRM; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-4.53 to 5.78] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 12: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 16; Test type: Other; MMRM; Mean Difference (Final Values) = 1.11, 95% CI 2-sided [-4.60 to 6.82] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 13: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 20; Test type: Other; MMRM; Mean Difference (Final Values) = 5.69, 95% CI 2-sided [-0.66 to 12.04] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 14: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 24; Test type: Other; MMRM; Mean Difference (Final Values) = 3.53, 95% CI 2-sided [-3.53 to 10.59] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)

5. Secondary Outcome: Change From Baseline in EuroQual 5 Dimensions (EQ-5D) VAS Score Over Time
Description: EQ-5D is a standardized instrument that measures the health-related quality of life. The EQ-5D consists of a descriptive system and a visual analog scale (VAS).The EQ-5D VAS records the patient's self-rated health on a vertical visual analogue scale with 0 representing 'Worst imaginable Health State' and 100 'Best imaginable Health State'. A positive change from baseline is a favorable outcome.
  The baseline value is defined as the last assessment performed prior to administration of the first dose of study treatment.
  A mixed effect model for repeated measurements (MMRM) was fitted to the changes from baseline in EQ-5D VAS score for all post-baseline time points up to Week 24. Values estimated from the model are presented in this table.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20 and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Remibrutinib 100 mg qd | Remibrutinib 100 mg Bid | Any Remibrutinib | Placebo
Number analyzed (Participants) | 24 | 23 | 47 | 23
score on scale
  Week 2 | -3.05 (3.11) | -2.86 (3.16) | -2.95 (2.22) | -3.02 (3.28)
  Week 4 | -1.74 (2.71) | -0.03 (2.86) | -0.88 (1.97) | 2.99 (2.87)
  Week 8 | 1.46 (3.20) | 1.76 (3.20) | 1.61 (2.26) | 3.44 (3.04)
  Week 12 | -2.36 (2.71) | 1.58 (2.82) | -0.39 (1.95) | 4.00 (2.64)
  Week 16 | -0.44 (3.27) | 4.27 (3.54) | 1.92 (2.41) | 1.79 (3.28)
  Week 20 | -0.91 (3.15) | 5.37 (3.33) | 2.23 (2.29) | 5.29 (3.01)
  Week 24 | 1.81 (3.47) | 5.73 (3.65) | 3.77 (2.52) | 2.07 (3.22)
Statistical Analysis 1: Comparison: Any Remibrutinib vs Placebo; Week 2; Test type: Superiority; p = 0.494, MMRM — one-sided p-value; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-7.84 to 7.96] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 2: Comparison: Any Remibrutinib vs Placebo; Week 4; Test type: Superiority; p = 0.866, MMRM — one-sided p-value; Mean Difference (Final Values) = -3.87, 95% CI 2-sided [-10.81 to 3.06] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 3: Comparison: Any Remibrutinib vs Placebo; Week 8; Test type: Superiority; p = 0.684, MMRM — one-sided p-value; Mean Difference (Final Values) = -1.82, 95% CI 2-sided [-9.37 to 5.73] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 4: Comparison: Any Remibrutinib vs Placebo; Week 12; Test type: Superiority; p = 0.908, MMRM — one-sided p-value; Mean Difference (Final Values) = -4.39, 95% CI 2-sided [-10.93 to 2.14] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 5: Comparison: Any Remibrutinib vs Placebo; Week 16; Test type: Superiority; p = 0.487, MMRM — one-sided p-value; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-8.00 to 8.26] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 6: Comparison: Any Remibrutinib vs Placebo; Week 20; Test type: Superiority; p = 0.790, MMRM — one-sided p-value; Mean Difference (Final Values) = -3.06, 95% CI 2-sided [-10.61 to 4.49]; Difference (Any remibrutinib - Placebo)
Statistical Analysis 7: Comparison: Any Remibrutinib vs Placebo; Week 24; Test type: Superiority; p = 0.340, MMRM — one-sided p-value; Mean Difference (Final Values) = 1.70, 95% CI 2-sided [-6.48 to 9.88] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 8: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 2; Test type: Other; MMRM; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-9.06 to 8.68] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 9: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 4; Test type: Other; MMRM; Mean Difference (Final Values) = -1.71, 95% CI 2-sided [-9.59 to 6.17] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 10: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 8; Test type: Other; MMRM; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-9.34 to 8.74] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 11: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 12; Test type: Other; MMRM; Mean Difference (Final Values) = -3.94, 95% CI 2-sided [-11.74 to 3.86] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 12: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 16; Test type: Other; MMRM; Mean Difference (Final Values) = -4.71, 95% CI 2-sided [-14.34 to 4.93] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 13: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 20; Test type: Other; MMRM; Mean Difference (Final Values) = -6.29, 95% CI 2-sided [-15.44 to 2.87] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 14: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 24; Test type: Other; MMRM; Mean Difference (Final Values) = -3.92, 95% CI 2-sided [-14.01 to 6.16] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)

6. Secondary Outcome: Change From Baseline in Physician Global Assessment Scale (PhGA) Score Over Time
Description: The physician's global assessment scale was used for the Investigator to rate the disease activity of their patient using 100 mm visual analog scale (VAS) ranging from "no disease activity" (0) to "maximal disease activity" (100). A negative change from baseline indicates improvement.
  The baseline value is defined as the last assessment performed prior to administration of the first dose of study treatment.
  A mixed effect model for repeated measurements (MMRM) was fitted to the changes from baseline in PhGA score for all post-baseline time points up to Week 24. Values estimated from the model are presented in this table.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20 and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Remibrutinib 100 mg qd | Remibrutinib 100 mg Bid | Any Remibrutinib | Placebo
Number analyzed (Participants) | 24 | 24 | 48 | 24
score on scale
  Week 2 | -4.21 (2.90) | -4.02 (2.85) | -4.12 (2.04) | -4.82 (3.10)
  Week 4 | -9.58 (2.89) | -8.93 (2.96) | -9.26 (2.08) | -7.28 (2.95)
  Week 8 | -13.68 (3.39) | -13.78 (3.28) | -13.73 (2.37) | -13.23 (3.16)
  Week 12 | -13.85 (3.63) | -9.45 (3.68) | -11.65 (2.60) | -17.67 (3.52)
  Week 16 | -19.37 (3.61) | -7.25 (3.74) | -13.31 (2.61) | -15.90 (3.51)
  Week 20 | -23.56 (3.43) | -17.31 (3.48) | -20.43 (2.45) | -17.57 (3.20)
  Week 24 | -21.25 (3.88) | -13.15 (3.95) | -17.20 (2.78) | -20.15 (3.54)
Statistical Analysis 1: Comparison: Any Remibrutinib vs Placebo; Week 2; Test type: Superiority; p = 0.575, MMRM — one-sided p-value; Mean Difference (Final Values) = 0.71, 95% CI 2-sided [-6.75 to 8.16] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 2: Comparison: Any Remibrutinib vs Placebo; Week 4; Test type: Superiority; p = 0.294, MMRM — one-sided p-value; Mean Difference (Final Values) = -1.98, 95% CI 2-sided [-9.22 to 5.27] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 3: Comparison: Any Remibrutinib vs Placebo; Week 8; Test type: Superiority; p = 0.450, MMRM — one-sided p-value; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-8.40 to 7.41] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 4: Comparison: Any Remibrutinib vs Placebo; Week 12; Test type: Superiority; p = 0.913, MMRM — one-sided p-value; Mean Difference (Final Values) = 6.02, 95% CI 2-sided [-2.74 to 14.78] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 5: Comparison: Any Remibrutinib vs Placebo; Week 16; Test type: Superiority; p = 0.722, MMRM — one-sided p-value; Mean Difference (Final Values) = 2.59, 95% CI 2-sided [-6.16 to 11.34] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 6: Comparison: Any Remibrutinib vs Placebo; Week 20; Test type: Superiority; p = 0.241, MMRM — one-sided p-value; Mean Difference (Final Values) = -2.86, 95% CI 2-sided [-10.96 to 5.24]; Difference (Any remibrutinib - Placebo)
Statistical Analysis 7: Comparison: Any Remibrutinib vs Placebo; Week 24; Test type: Superiority; p = 0.742, MMRM — one-sided p-value; Mean Difference (Final Values) = 2.95, 95% CI 2-sided [-6.09 to 11.99] — Difference (Any remibrutinib - Placebo)
Statistical Analysis 8: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 2; Test type: Other; MMRM; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-8.28 to 7.91] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 9: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 4; Test type: Other; MMRM; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-8.87 to 7.58] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 10: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 8; Test type: Other; MMRM; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-9.28 to 9.48] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 11: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 12; Test type: Other; MMRM; Mean Difference (Final Values) = -4.40, 95% CI 2-sided [-14.71 to 5.90] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 12: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 16; Test type: Other; MMRM; Mean Difference (Final Values) = -12.1, 95% CI 2-sided [-22.47 to -1.77] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 13: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 20; Test type: Other; MMRM; Mean Difference (Final Values) = -6.25, 95% CI 2-sided [-16.00 to 3.50] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)
Statistical Analysis 14: Comparison: Remibrutinib 100 mg qd vs Remibrutinib 100 mg Bid; Week 24; Test type: Other; MMRM; Mean Difference (Final Values) = -8.10, 95% CI 2-sided [-19.16 to 2.96] — Difference (remibrutinib 100 mg qd - remibrutinib 100 mg bid)

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: Number of participants with TEAEs and serious TEAEs, including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as TEAEs. TEAEs are defined as adverse events that started after the first dose of study medications or adverse events present prior to start of double-blind treatment but increased in severity.
  The number of participants in each category is reported in the table.
Time Frame: From first dose of study treatment up 30 days after last dose (Week 29)
Population: Safety Analysis Set defined as participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Remibrutinib 100 mg Bid | Remibrutinib 100 mg qd | Placebo
Number analyzed (Participants) | 24 | 25 | 24
Participants
  TEAE | 22 | 21 | 20
  Study drug-related TEAE | 10 | 8 | 9
  Serious TEAE | 1 | 1 | 1

8. Secondary Outcome: Maximum Observed Blood Concentration (Cmax) of Remibrutinib at Week 4
Description: Remibrutinib was determined in whole blood by a validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) method with a lower limit of quantification (LLOQ) of 1.0 ng/mL. Pharmacokinetic (PK) parameters were calculated based on remibrutinib blood concentrations by using the actual recorded sampling times and non-compartmental methods with Phoenix WinNonlin (version 8 or higher). Concentrations below the LLOQ were treated as zero. Cmax is defined as the maximum (peak) observed blood concentration following a dose.
Time Frame: pre-dose, 0.5, 1, 2, 3 and 4 hours post-dose at Week 4
Population: Participants in the PK Analysis Set (PKS) with a valid value for the outcome measure. PKS is defined as participants with at least one available valid PK concentration measurement, who received any study drug, and with no protocol deviations that impact PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Remibrutinib 100 mg Bid | Remibrutinib 100 mg qd
Number analyzed (Participants) | 16 | 13
ng/mL | 183 (82.5) | 225 (154)

9. Secondary Outcome: Maximum Observed Blood Concentration (Cmax) of Remibrutinib at Week 24
Description: as for outcome 8
Time Frame: pre-dose, 0.5, 1, 2, 3 and 4 hours post-dose at Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Remibrutinib 100 mg Bid | Remibrutinib 100 mg qd
Number analyzed (Participants) | 14 | 10
ng/mL | 224 (202) | 169 (77.9)

10. Secondary Outcome: Time to Reach Maximum Observed Blood Concentration (Tmax) of Remibrutinib at Week 4
Description: Remibrutinib was determined in whole blood by a validated LC-MS/MS method with a LLOQ of 1.0 ng/mL. Pharmacokinetic (PK) parameters were calculated based on remibrutinib blood concentrations by using the actual recorded sampling times and non-compartmental methods with Phoenix WinNonlin (version 8 or higher). Concentrations below the LLOQ were treated as zero. Tmax is defined as the time to reach maximum (peak) blood concentration following a dose.
Time Frame: pre-dose, 0.5, 1, 2, 3 and 4 hours post-dose at Week 4
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Remibrutinib 100 mg Bid | Remibrutinib 100 mg qd
Number analyzed (Participants) | 16 | 13
hours | 1.00 [0.500 to 3.00] | 1.00 [0.500 to 4.00]

11. Secondary Outcome: Time to Reach Maximum Observed Blood Concentration (Tmax) of Remibrutinib at Week 24
Description: as for outcome 10
Time Frame: pre-dose, 0.5, 1, 2, 3 and 4 hours post-dose at Week 24
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Remibrutinib 100 mg Bid | Remibrutinib 100 mg qd
Number analyzed (Participants) | 14 | 10
hours | 1.00 [0.500 to 3.00] | 1.00 [0.500 to 3.08]

12. Secondary Outcome: Area Under the Blood Concentration-time Curve Within a Dosing Interval (Tau) at Steady-state (AUCtau) of Remibrutinib at Week 4
Description: Remibrutinib was determined in whole blood by a validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) method with a lower limit of quantification (LLOQ) of 1.0 ng/mL. Pharmacokinetic (PK) parameters were calculated based on remibrutinib blood concentrations by using the actual recorded sampling times and non-compartmental methods with Phoenix WinNonlin (version 8 or higher). Concentrations below the LLOQ were treated as zero. AUCtau is defined as the area under the blood concentration-time curve calculated/extrapolated to the end of a dosing interval (tau) at steady-state. Tau was 24 hours for the qd dosing group and 12 hours for the bid dosing group. For the calculation of AUCtau, the pre-dose concentrations at Week 4 and Week 24 were duplicated as 24 hours and 12 hours concentrations for the qd and bid groups, respectively. The linear trapezoidal method was used for AUCtau calculation.
Time Frame: pre-dose, 0.5, 1, 2, 3 and 4 hours post-dose at Week 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Remibrutinib 100 mg Bid | Remibrutinib 100 mg qd
Number analyzed (Participants) | 16 | 8
h*ng/mL | 569 (311) | 1020 (700)

13. Secondary Outcome: Area Under the Blood Concentration-time Curve Within a Dosing Interval (Tau) at Steady-state (AUCtau) of Remibrutinib at Week 24
Description: as for outcome 12
Time Frame: pre-dose, 0.5, 1, 2, 3 and 4 hours post-dose at Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Remibrutinib 100 mg Bid | Remibrutinib 100 mg qd
Number analyzed (Participants) | 14 | 6
h*ng/mL | 670 (380) | 636 (306)

14. Secondary Outcome: Area Under the Blood Concentration-time Curve From Time Zero to 4 Hours Post-dose (AUC0-4h) of Remibrutinib at Week 4
Description: Remibrutinib was determined in whole blood by a validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) method with a lower limit of quantification (LLOQ) of 1.0 ng/mL. Pharmacokinetic (PK) parameters were calculated based on remibrutinib blood concentrations by using the actual recorded sampling times and non-compartmental methods with Phoenix WinNonlin (version 8 or higher). Concentrations below the LLOQ were treated as zero. AUC0-4h is defined as the area under the blood concentration-time curve from time zero to 4 hours post-dose, which was the last sampling time. The linear trapezoidal method was used for AUC0-4h calculation.
Time Frame: pre-dose, 0.5, 1, 2, 3 and 4 hours post-dose at Week 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Remibrutinib 100 mg Bid | Remibrutinib 100 mg qd
Number analyzed (Participants) | 16 | 13
h*ng/mL | 351 (169) | 393 (207)

15. Secondary Outcome: Area Under the Blood Concentration-time Curve From Time Zero to 4 Hours Post-dose (AUC0-4h) of Remibrutinib at Week 24
Description: as for outcome 14
Time Frame: pre-dose, 0.5, 1, 2, 3 and 4 hours post-dose at Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Remibrutinib 100 mg Bid | Remibrutinib 100 mg qd
Number analyzed (Participants) | 14 | 10
h*ng/mL | 420 (259) | 317 (144)

16. Secondary Outcome: Elimination Half-life (T1/2) of Remibrutinib at Week 4
Description: Remibrutinib was determined in whole blood by a validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) method with a lower limit of quantification (LLOQ) of 1.0 ng/mL. Pharmacokinetic (PK) parameters were calculated based on remibrutinib blood concentrations by using the actual recorded sampling times and non-compartmental methods with Phoenix WinNonlin (version 8 or higher). Concentrations below the LLOQ were treated as zero. T1/2 is defined as the time taken for the blood concentration, as well as the amount of the drug in the body, to fall by one-half.
Time Frame: pre-dose, 0.5, 1, 2, 3 and 4 hours post-dose at Week 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Remibrutinib 100 mg Bid | Remibrutinib 100 mg qd
Number analyzed (Participants) | 11 | 9
hours | 3.08 (0.998) | 3.86 (2.28)

17. Secondary Outcome: Elimination Half-life (T1/2) of Remibrutinib at Week 24
Description: as for outcome 16
Time Frame: pre-dose, 0.5, 1, 2, 3 and 4 hours post-dose at Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Remibrutinib 100 mg Bid | Remibrutinib 100 mg qd
Number analyzed (Participants) | 11 | 8
hours | 3.15 (0.907) | 3.88 (1.95)

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up 30 days after last dose (Week 29)
Description: Any sign or symptom that occurs from first dose of study treatment up to 30 days after last dose.
Groups:
- Remibrutinib 100 mg qd: Remibrutinib 100 mg qd
- Total: All participants
Arm/Group | Remibrutinib 100 mg Bid | Remibrutinib 100 mg qd | Any Remibrutinib | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25 | 0/49 | 0/24 | 0/73
Serious Adverse Events (participants affected / at risk) | 1/24 | 1/25 | 2/49 | 1/24 | 3/73
Other Adverse Events (participants affected / at risk) | 15/24 | 12/25 | 27/49 | 17/24 | 44/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remibrutinib 100 mg Bid (N=24) | Remibrutinib 100 mg qd (N=25) | Any Remibrutinib (N=49) | Placebo (N=24) | Total (N=73)
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remibrutinib 100 mg Bid (N=24) | Remibrutinib 100 mg qd (N=25) | Any Remibrutinib (N=49) | Placebo (N=24) | Total (N=73)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 2 | 4
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 1 | 3
Nausea (Gastrointestinal disorders) | 4 | 1 | 5 | 2 | 7
Asthenia (General disorders) | 0 | 2 | 2 | 1 | 3
Fatigue (General disorders) | 3 | 0 | 3 | 2 | 5
Nasopharyngitis (Infections and infestations) | 2 | 1 | 3 | 3 | 6
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 3 | 2 | 5
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 2 | 4
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0 | 2
Blood immunoglobulin G increased (Investigations) | 0 | 0 | 0 | 2 | 2
White blood cell count decreased (Investigations) | 2 | 1 | 3 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 2 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 3
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 2
Headache (Nervous system disorders) | 1 | 3 | 4 | 5 | 9
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT04035668/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT04035668/SAP_001.pdf